CLINICAL TRIAL: NCT02426346
Title: TEEN JOIN: A Scalable Weight Control Intervention for Adolescents
Brief Title: A Scalable Weight Control Intervention for Adolescents
Acronym: TEEN JOIN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Elissa Jelalian, Associate Professor, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34DK10098101A1
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Pediatric Obesity
Keywords: Adolescent; Adolescent obesity; Community-based; Overweight
MeSH Terms: conditions — Pediatric Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JOIN FOR ME (Active Comparator): The JOIN for ME curriculum includes 16 weekly in person sessions followed by 4 biweekly and 4 monthly maintenance sessions for a 10-month program. Weekly meetings are scheduled for 60 minutes and are facilitated by a YMCA coach. Interventions include behavioral weight control and parent-based incentives. Parents attend group at weeks 1, 2 and 16 with their teen.
  Interventions: Behavioral: Behavioral weight control; Behavioral: Parent-based incentives
- TEEN JOIN (Experimental): Similar to the JOIN FOR ME condition, adolescents in the TEEN JOIN condition attend 16 weekly in person sessions followed by 4 biweekly and 4 monthly maintenance sessions for a 10-month program. Interventions include behavioral weight control, group-based physical activity, and group-based incentives. Parents attend separate meetings at weeks 1, 2, and 16.
  Interventions: Behavioral: Behavioral weight control; Behavioral: Group-based physical activity; Behavioral: Group-based incentives

INTERVENTIONS:
Behavioral: Behavioral weight control — Prescription of diet & physical activity and behavioral strategies for weight control
Behavioral: Group-based physical activity — Teens exercise for 60 minutes with their group
  Arms: TEEN JOIN
Behavioral: Group-based incentives — Adolescents earn reinforcements within group
  Arms: TEEN JOIN
Behavioral: Parent-based incentives — Adolescents earn reinforcements from their parents (outside of group)
  Arms: JOIN FOR ME

SUMMARY:
Community-based programs are needed to improve dissemination of efficacious treatment for adolescent obesity. The current study aims to modify a community-based program, delivered through the YMCA, to increase its effectiveness with adolescents. Adolescents will be randomized to either a 16-week standard program (JOIN) or a targeted intervention tailored for adolescents (TEEN JOIN). Primary outcomes include changes in BMI, objectively measured physical activity, and self-efficacy, assessed at 4 months and 10 months following randomization.

DETAILED DESCRIPTION:
In 2010, the U.S. Preventive Services Task Force (USPSTF) provided a Grade recommendation B (i.e. the service is recommended with moderate/high certainty of benefit) for clinicians to screen children ages 6-17 years for obesity and refer identified youth to comprehensive behavioral programs. The challenge in meeting this objective is the lack of community-based obesity treatments to which to refer, particularly for adolescents. The JOIN program, developed as a collaboration between United HealthGroup and Y-USA is a pediatric weight control intervention targeted toward a broad age range of youth from 6-17 years that is: 1) based on well established and evidence based principles; 2) delivered by YMCA facilitators within a community setting: and 3) potentially scalable nationally. Findings from a 6-month pilot study examining the effectiveness of JOIN demonstrated impressive changes in weight status for school age children, but more modest results for adolescents. The primary aim of this study is to modify the JOIN program to increase its effectiveness with adolescents while retaining its potential for scalability.

A total of 120 adolescents (ages 13-17) with BMI > 85th% and < 50 will be randomly assigned to a 16-week targeted program (TEEN JOIN), or the traditional JOIN intervention, followed by biweekly and monthly maintenance sessions. Evaluation of adolescent height, weight, objective physical activity and psychosocial outcomes will be obtained at baseline, 4 months, and 10 months. Additional outcomes will include treatment feasibility, including attendance, completion of diet and physical activity monitoring logs, and exit interviews with adolescents and parents regarding the intervention. The investigators will also obtain preliminary indicators of cost effectiveness. It is hypothesized that adolescents who are randomized to TEEN JOIN will demonstrate greater decrease in BMI at 4 and 10 months than those randomized to JOIN. It is further hypothesized that adolescents randomized to TEEN JOIN will demonstrate greater increases in participation in moderate-vigorous physical activity and greater improvements in self-concept, self-efficacy related to physical activity, and group cohesion than adolescents who receive the standard JOIN condition.

ELIGIBILITY:
Inclusion Criteria:

* 13 to 17 years
* BMI > 85th percentile and absolute BMI < 50
* have at least one parent available to provide consent and participate in sessions
* speak English
* agree to study participation and random assignment

Exclusion Criteria:

* currently involved in another weight loss program
* have a medical condition that would interfere with the prescribed dietary plan or participation in physical activity
* developmentally delayed such that the intervention materials will not be appropriate
* in treatment for a major psychiatric disorder, including an eating disorder, or are diagnosed with a major psychiatric disorder at the time of screening.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI, kg/m2) | Baseline, post-treatment 1 (4 months), post-treatment 2 (10 months)

SECONDARY OUTCOMES:
Objective time spent in moderate and vigorous physical activity measured by the Senswear Mini (MINI) armband | Baseline, post-treatment 1 (4 months), post-treatment 2 (10 months)
  Objectively-measured moderate and vigorous physical activity
Self-Efficacy Questionnaire | Baseline, post-treatment 1 (4 months), post-treatment 2 (10 months)
  Adolescents' confidence in their ability to lose weight and engage in physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- Weight Management and Diabetes Research Center, The Miriam Hospital/Alpert Medical School of Brown University, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Jelalian E, Evans EW, Rancourt D, Ranzenhofer L, Taylor N, Hart C, Seifer R, Klinepier K, Foster GD. JOIN for ME: Testing a Scalable Weight Control Intervention for Adolescents. Child Obes. 2020 Apr;16(3):192-203. doi: 10.1089/chi.2019.0053. Epub 2019 Dec 18. PMID 31855057